CLINICAL TRIAL: NCT02448771
Title: A Phase Ib/II Study of Palbociclib in Combination With Bazedoxifene in Hormone Receptor Positive Breast Cancer
Brief Title: A Study of Palbociclib in Combination With Bazedoxifene in Hormone Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Rinath Jeselsohn MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-060
Record Dates: First submitted 2015-05-04; First posted 2015-05-19 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Stage IV; Unresectable Locally Advanced Invasive Breast Cancer; Metastatic Invasive Breast Cancer
Keywords: Unresectable locally advanced invasive breast cancer; Metastatic invasive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; bazedoxifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palbociclib in Combination with Bazedoxifene (Experimental): Palbociclib 125 mg Oral on days 1-21 per cycle Bazedoxifene 40 mg Oral on days 1-28 per cycle
  One cycle is 28 days.
  Interventions: Drug: Palbociclib; Drug: Bazedoxifene

INTERVENTIONS:
Drug: Palbociclib
  Other Names: Ibrance
Drug: Bazedoxifene
  Other Names: TSE-424 (IS); UNII-Q16TT9C5BK (IS); WAY 140424 (IS)

SUMMARY:
This research study is studying a drug called Palbociclib in combination with Bazedoxifene (a type of endocrine therapy, which prevents breast cancer cell growth by blocking estrogen stimulation) as a possible treatment for this diagnosis.

The names of the study interventions involved in this study are:

* Palbociclib
* Bazedoxifene

DETAILED DESCRIPTION:
This research study is a Phase I/II clinical trial. Phase II clinical trial tests the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved Palbociclib in combination with Bazedoxifene for use in participants with your type of cancer, but it has been approved for other uses (metastatic breast cancer).

Palbociclib is a drug that may stop cancer cells from growing. Palbociclib blocks activity of two closely related enzymes (proteins that help chemical reactions in the body occur), called Cyclin D Kinases 4 and 6 (CDK 4/6). These proteins are part of a pathway, or a sequence of steps which is known to control cell growth. Laboratory testing has shown that palbociclib may stop the growth of hormone receptor positive breast cancer.

Endocrine therapy prevents breast cancer cell growth by blocking the activity of the estrogen receptor. During this study the endocrine therapy will be bazedoxifene.

In this research study, the investigators are evaluating how safe palbociclib is and how well palbociclib in combination with bazedoxifene, a form of endocrine treatment, works in participants with a history of stage four breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed invasive breast cancer that is metastatic or unresectable locally advanced. Histological documentation of metastatic/recurrent breast cancer is not required if there is unequivocal evidence for recurrence of the breast cancer.
* Estrogen and/or progesterone receptor positive breast cancer (>10% staining), as determined by pathology from either primary or metastatic site(s). Central confirmation is not required.
* HER2 negative, defined as 0-1+ by immunohistochemistry or FISH-negative (HER2 copy number <6 and HER2/CEP17 ratio < 2.0). Central confirmation is not required.
* Postmenopausal women are eligible. Postmenopausal is defined as any of the following:

  * Age ≥60 years
  * Age <60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifen, or ovarian suppression) and FSH and estradiol in the postmenopausal range per local normal range.
  * Premenopausal women who have been on a GnRH agonist for at least 3 consecutive months prior to study entry are eligible. Women in this group MUST remain on the GnRH agonist for the duration of protocol treatment.
  * Status-post bilateral oophorectomy-After adequate healing post surgery.
  * Women, age ≥18 years of age. Men are excluded.
  * Because no dosing or adverse event data are currently available on the use of palbociclib and bazedoxifene in participants <18 years of age, children are excluded from this study. In addition, breast cancer is exceedingly rare in individuals under 18 years of age.
* Participants must have measurable disease by RECIST 1.1. See section 11 for the definition of measurable disease.
* Bone only disease if there are lytic lesions is also allowed and treatment response will be evaluated based on the MD Anderson criteria. See section 11.
* Endocrine resistant breast cancer, defined as either:

  * Relapsed while on adjuvant endocrine therapy or within 1 year of completion of adjuvant endocrine therapy

    --- -or-
  * Progression through at least one line of endocrine therapy for metastatic or locally advanced breast cancer. There is no limit on the number of prior endocrine therapies received.
  * Patients may have received up to one prior line of chemotherapy for metastatic or unresectable locally advanced breast cancer.
  * Patients may have initiated bisphosphonate therapy prior to start of protocol therapy. Bisphosphonate therapy may continue during protocol treatment. Such patients will have bone lesions considered evaluable for progression
  * Patients must be at least 2 weeks from prior chemotherapy or radiotherapy, or any investigational drug product, with adequate recovery of toxicity to baseline, or grade <1, with the exception of alopecia and hot flashes. There is no washout period for prior endocrine therapy.
* ECOG Performance Status 0-1 (Appendix A)
* Life expectancy of greater than 3 months
* Willingness to undergo research biopsy under the following circumstances:

  * Patients with "easily accessible disease"

    * Patients with skin or chest wall disease amenable to a punch biopsy under local anesthesia are required to undergo a baseline biopsy and a biopsy at the time of disease progression as part of this protocol.
    * Patients with a breast mass or axillary lymph node amenable to an image-guided core biopsy are also required to undergo a baseline biopsy and a biopsy at the time of disease progression as part of this protocol.
    * Patients with malignant ascites fluid or a malignant pleural effusion of sufficient volume to be amenable to tap (either in-office or image-guided) are also required to undergo a baseline tap and a tap at the time of disease progression as part of this protocol.
    * Patients who undergo a research biopsy procedure for the purpose of this protocol, and in whom inadequate tissue is obtained, are still eligible and are not required to undergo a repeat biopsy in order to enter the study.
    * Patients will be approached during cycle 1 about providing an optional tissue sample at that time; however, this biopsy will be optional.
  * Patients with "accessible disease"

    * Patients with sites felt to be accessible to an image-guided or incisional biopsy in the opinion of the patient's treating oncologist and physician performing the procedure, and not meeting the criteria for "easily accessible disease" as described in Section 3.1.14.1, are required to undergo a baseline biopsy as part of this protocol. Such sites may include, but are not limited to: liver, lymph nodes, soft tissue, lung, chest wall, and bone. Cycle 1 biopsy and biopsy at time of disease progression are optional.
    * Biopsies may be done with local anesthesia or intravenous conscious sedation, according to standard institutional guidelines.
    * If a biopsy requires general anesthesia, then it is only allowed if acquisition of tissue is necessary for clinical reasons (i.e. is clinically indicated), and excess tissue that would otherwise have been discarded is then used for research purposes. If a biopsy requires general anesthesia, then a biopsy of that site for research purposes only, without a coexisting clinical indication is not allowed on this protocol.
    * Patients who undergo a research biopsy procedure for the purpose of this protocol, and in whom inadequate tissue is obtained, are still eligible and are not required to undergo a repeat biopsy in order to enter the study.
    * Some patients may have had a clinically indicated biopsy upon recent disease progression. No additional pre-treatment biopsy is required if that specimen can be used for the correlative studies described in this protocol.
    * Patients will be approached at the time of progression about providing an optional tissue sample at that time; however, the time of progression biopsy will be optional.
  * Other patients

    * Patients who do not have biopsy-accessible disease are not required to undergo a biopsy as part of study participation.
    * In addition, patients who are being treated with therapeutic doses of anticoagulant(s), are not required to undergo a biopsy as part of study participation. If it is felt clinically appropriate despite anticoagulation (i.e. a skin punch biopsy, etc) by the treating physician, a biopsy is allowed, it is simply not required.
    * The sites of metastatic disease and reason that the disease is not biopsy-accessible should be documented in the medical record and case report form(s).
    * Patients who do not undergo baseline biopsy must have their study participation approved by the overall PI before start of protocol therapy. Only patients who have biopsy inaccessible disease may enter the study without the requirement for baseline biopsy.
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Hgb ≥9 mg/dL (which may be post transfusion)
  * Total bilirubin ≤1.5 X institutional upper limit of normal (patients with

    ---- documented Gilbert's disease are allowed total bilirubin up to 3X ULN)
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit if no liver metastases; and ≤ 5 X institutional upper limit if liver metastases are present.
  * Creatinine ≤ 2X institutional upper limit of normal
  * Baseline QTc ≤ 480 ms
* Ability to take oral medications.
* The effects of palbociclib and bazedoxifene on the developing human fetus are unknown. If, for any reason, a woman should become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.
* Women who are made postmenopausal through use of GNRH agonists, and men are required to use adequate contraception for the duration of protocol treatment and for 6 months after the last dose of palbociclib and bazedoxifene. Adequate contraception is defined as one highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the patient and/or partner.
* Highly Effective Non-Hormonal Contraception Methods of birth control which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly are considered highly-effective forms of contraception. The following non-hormonal methods of contraception are acceptable:

  * True abstinence when this is in line with the preferred and usual lifestyle of the patient. [Periodic abstinence (e.g., calendar, ovulation, symptothermal post-ovulation methods) and withdrawal are not acceptable methods of contraception].
  * Male sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female patients, the vasectomized male partner should be the sole partner.

    --- OR
  * Effective Non-Hormonal Contraception

Alternatively two of the following effective forms of contraception may be used instead:

* Placement of non-hormonal intrauterine device (IUD) or intrauterine system (IUS). Consideration should be given to the type of device being used, as there is higher failure rates quoted for certain types, e.g., steel or copper wire.
* Condom with spermicidal foam/gel/film/cream/suppository.
* Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository. The use of barrier contraceptives should always be supplemented with the use of spermicide.

  - The following should be noted:
* Failure rates indicate that, when used alone, the diaphragm and ondom are not highly effective forms of contraception. Therefore, the use of additional spermicides does confer additional theoretical contraceptive protection.
* However, spermicides alone are ineffective at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

  * It should be noted that two forms of effective contraception are required. A double barrier method is acceptable, which is defined as condom and occlusive cap (diaphragm or cervical/ vault caps) with spermicidal foam/gel/film/cream /suppository. Premenopausal women who have been on a GnRH agonist for at least 3 consecutive months prior to study entry are eligible. Women in this group MUST remain on the GnRH agonist for the duration of protocol treatment. Such patients should be counseled that GnRH agonists alone may not be adequate contraception and that adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation should be employed.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with a CDK4/6 inhibitor and/or bazedoxifene.
* Participants may not be receiving any other investigational agents.
* Concurrent treatment with commercial agents or other agents with the intent to treat the participant's malignancy, including endocrine therapy, chemotherapy, and/or targeted therapy, with the exception of bisphosphonates and GnRH agonists, as detailed in sections 3.1.4 and 3.1.9.
* Untreated or progressive brain metastases. Patients with treated brain metastases not requiring chronic corticosteroids for symptom control are eligible.
* Pending visceral crisis, in the opinion of the treating investigator.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib and /or bazedoxifene.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A isoenzymes are ineligible. Lists including medications and substances known or with the potential to interact with the CYP3A isoenzymes are provided in Appendix D. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Current use of drugs that are known to prolong the QT interval (See Appendix C)
* Subjects with organ allograft requiring immunosuppression.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Ability to comply with study requirements is to be assessed by each investigator at the time of screening for study participation.
* Pregnant women are excluded from this study because effects of palbociclib and bazedoxifene on a developing fetus is unknown. Breastfeeding should be discontinued prior to entry onto the study.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Patients on combination antiretroviral therapy, i.e. those who are HIV-positive, are ineligible because of the potential for pharmacokinetic interactions or significant immunosuppression with Palbociclib.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rinath Jelsohn, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Tsuji J, Li T, Grinshpun A, Coorens T, Russo D, Anderson L, Rees R, Nardone A, Patterson C, Lennon NJ, Cibulskis C, Leshchiner I, Tayob N, Tolaney SM, Tung N, McDonnell DP, Krop IE, Winer EP, Stewart C, Getz G, Jeselsohn R. Clinical Efficacy and Whole-Exome Sequencing of Liquid Biopsies in a Phase IB/II Study of Bazedoxifene and Palbociclib in Advanced Hormone Receptor-Positive Breast Cancer. Clin Cancer Res. 2022 Dec 1;28(23):5066-5078. doi: 10.1158/1078-0432.CCR-22-2305. PMID 36215125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 7/9/2015 and 7/19/2017
Period: Overall Study
Arm/Group | Palbociclib in Combination With Bazedoxifene
Started | 36
Completed | 0
Not Completed | 36
Not completed — Disease Progression | 30
Not completed — Unacceptable Toxicity | 1
Not completed — Physician Decision | 3
Not completed — Started new therapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 59.5 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 1
  Unknown or Not Reported | 3
ECOG Performance Status [Count of Participants; unit: Participants]
  00 - Fully Active | 33
  01 - Restricted | 3
Estrogen Receptor Status [Count of Participants; unit: Participants]
  Unknown | 1
  Low Positive | 1
  Positive (>10% cell staining) | 34
Progesterone Receptor Status [Count of Participants; unit: Participants]
  Unknown | 1
  Low Positive | 1
  Positive (>10% cell staining) | 22
  Negative (<=10% cell staining) | 12
Human Epidermal Growth Factor Receptor 2 Amplification [Count of Participants; unit: Participants]
  Negative | 36
  Positive | 0
Site of Metastatic Disease [Count of Participants; unit: Participants]
  Lung and Pleural | 12
  Breast and Chest | 14
  Lymph Node | 13
  Liver | 23
  Bone | 26
  Others | 7
Site of Metastatic Disease: Bone Only [Count of Participants; unit: Participants]
  Yes | 2
  No | 34
Site of Metastatic Disease: Visceral Disease [Count of Participants; unit: Participants]
  Yes | 29
  No | 7
Prior Hormonal Therapy for Metastatic Breast Cancer [Count of Participants; unit: Participants]
  Zero | 6
  One | 14
  Two | 8
  Three | 6
  Four | 2
Prior Chemotherapy for Metastatic Breast Cancer [Count of Participants; unit: Participants]
  Zero | 17
  One | 16
  Two | 3
Everolimus for Metastatic Breast Cancer [Count of Participants; unit: Participants]
  Yes | 4
  No | 32
Prior Hormonal Therapy for Primary Cancer [Count of Participants; unit: Participants]
  Yes | 25
  No | 11
Prior Tamoxifen for Primary or Metastatic Breast Cancer [Count of Participants; unit: Participants]
  Yes | 26
  No | 10

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: Clinical Benefit Rate is the percentage of participants who achieve clinical benefit from the study treatment. Clinical benefit is defined as at least 24 weeks of confirmed Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
  SD or better is achieved if the following are true:
  Target Lesions:
  -At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Non-target Lesions:
  * No progression.
  * No appearance new lesions or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
  Bone Lesions:
  * < 25% increase in lesions.
  * No new lesions.
Time Frame: Assessed for response for up to 34 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 36
percentage of participants | 33 [9.8 to 56.4]

2. Primary Outcome: Clinical Benefit Rate by ESR1 Genotype
Description: Clinical Benefit Rate is the percentage of participants who achieve clinical benefit from the study treatment. Clinical benefit is defined as at least 24 weeks of confirmed CR, PR, SD.
  SD or better is achieved if the following are true:
  Target Lesions:
  -At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Non-target Lesions:
  * No progression.
  * No appearance new lesions or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
  Bone Lesions:
  * < 25% increase in lesions.
  * No new lesions.
  ESR1 genotype determined using established methods
Time Frame: Assessed for response for up to 34 months
Population: Total number analyzed is the sum of both categories (mutant and wild type).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 28
percentage of participants
  Wild Type: number analyzed (Participants) | 16
  Wild Type | 31 [11.0 to 58.67]
  Mutant: number analyzed (Participants) | 7
  Mutant | 43 [9.9 to 81.6]

3. Primary Outcome: Percent of Participants With All Grade Neutrophil Count Decrease
Description: Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 regardless of whether the event is related or unrelated to treatment. Neutrophil counts are evaluated using established methods.
Time Frame: Baseline, until resolution or for 30 days after the subject's last study visit, up to 43 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Palbociclib in Combination With Bazedoxifene: Palbociclib 125 mg Oral on days 1-21 per cycle Bazedoxifene 40 mg Oral on days 1-28 per cycle
  One cycle is 28 days.
  Palbociclib
  Bazedoxifene
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 36
percentage of participants | 61.1 [45 to 77]

4. Secondary Outcome: Number of Participants With All Grade Neutrophil Count Decrease
Description: as for outcome 3
Time Frame: Baseline, until resolution or for 30 days after the subject's last study visit, up to 43 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 36
Participants | 22

5. Secondary Outcome: Objective Response Rate
Description: The objective response rate is the proportion of participants achieving complete response (CR) or partial response (PR) on treatment based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria.
  PR or better is achieved if the following are true:
  Target Lesions:
  -At least a 30% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Non-target Lesions:
  * No progression.
  * No appearance new lesions or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
  Bone Lesions:
  ->50% increase in lesions.
  -No new lesions.
Time Frame: Assessed for response for up to 34 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 36
percentage of participants | 11.1 [3.1 to 26.4]

6. Secondary Outcome: Median Progression-Free Survival
Description: Progression free survival (PFS) is defined as the time from start of treatment to disease progression or death from any cause as estimated by Kaplan Meier methods. Progression is measured using RECIST 1.1 criteria, defined as at least a 20% increase in size in target lesion and/or unequivocal progression of non-target lesions and/or appearance of new lesions. Patients who have not progressed and are alive are censored at the date the patient is known to be progression-free.
Time Frame: Up to 42 months
Population: Rows are representative of subgroups of study population.
Measure: Median (Full Range); unit: months
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 36
months | 3.58 [1.97 to 7.24]

7. Secondary Outcome: Median Overall Survival
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Time Frame: Up to 42 months
Measure: Median (Full Range); unit: months
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 36
months | 26.5 [1.5 to 41.5]

8. Secondary Outcome: Median Progression-Free Survival for Patients by ESR1 Genotype
Description: Progression free survival (PFS) is defined as the time from start of treatment to disease progression or death from any cause as estimated by Kaplan Meier methods. Patients who have not progressed and are alive are censored at the date the patient is known to be progression-free. ESR1 genotype is determined using established methods. Progression is measured using RECIST 1.1 criteria, defined as at least a 20% increase in size in target lesion and/or unequivocal progression of non-target lesions and/or appearance of new lesions
Time Frame: Up to 24 months
Population: Total number analyzed is the sum of both categories (mutant and wild type).
Measure: Median (Full Range); unit: months
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 27
months
  Mutant: number analyzed (Participants) | 10
  Mutant | 2.0 [1.5 to 9.3]
  Wild Type: number analyzed (Participants) | 17
  Wild Type | 3.6 [1.9 to 5.7]

9. Secondary Outcome: Overall Survival by ESR1 Genotype
Description: Overall Survival (OS) is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive. ESR1 genotype determined by established methods.
Time Frame: Up to 42 months
Population: Total number analyzed is the sum of both categories (mutant and wild type).
Measure: Median (95% Confidence Interval); unit: probability of survival
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 23
probability of survival
  Wild Type: number analyzed (Participants) | 16
  Wild Type | 21.1 [13.2 to NA] — Follow-up is not long enough/data is not mature to provide upper bound confidence interval.
  Mutant: number analyzed (Participants) | 7
  Mutant | 26.5 [1.5 to NA] — Follow-up is not long enough/data is not mature to provide upper bound confidence interval.

10. Secondary Outcome: Objective Response Rate by ESR1 Genotype
Description: The objective response rate is the proportion of participants achieving complete response (CR) or partial response (PR) on treatment based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria.
  PR or better is achieved if the following are true:
  Target Lesions:
  -At least a 30% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Non-target Lesions:
  No progression. No appearance new lesions or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
  Bone Lesions:
  ->50% increase in lesions.
  -No new lesions.
  ESR1 genotype determined by established methods.
Time Frame: Up to 34 months
Population: Total number analyzed is the sum of both categories (mutant and wild type).
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib in Combination With Bazedoxifene
Number analyzed (Participants) | 28
Participants
  Wild Type: number analyzed (Participants) | 19
  Wild Type: Complete Response | 0
  Wild Type: Partial Response | 0
  Wild Type: Stable Disease | 13
  Wild Type: Progressive Disease | 5
  Wild Type: Not Evaluable | 1
  Mutant: number analyzed (Participants) | 9
  Mutant: Complete Response | 0
  Mutant: Partial Response | 0
  Mutant: Stable Disease | 3
  Mutant: Progressive Disease | 5
  Mutant: Not Evaluable | 1

ADVERSE EVENTS:
Time Frame: Baseline, until resolution or for 30 days after the subject's last study visit, up to 43 months.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Palbociclib in Combination With Bazedoxifene
All-Cause Mortality (participants affected / at risk) | 17/36
Serious Adverse Events (participants affected / at risk) | 17/36
Other Adverse Events (participants affected / at risk) | 34/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib in Combination With Bazedoxifene (N=36)
Anemia (Blood and lymphatic system disorders) | 1
Bladder infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 15
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib in Combination With Bazedoxifene (N=36)
Anemia (Blood and lymphatic system disorders) | 6
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 12
Obstruction gastric (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 22
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 5
Lung infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 2
Rhinitis infective (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 3
Infections and infestations - Other, specify (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 5
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 21
Platelet count decreased (Investigations) | 8
Weight gain (Investigations) | 1
White blood cell decreased (Investigations) | 3
Investigations - Other, specify (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Movements involuntary (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urinary urgency (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Hot flashes (Vascular disorders) | 6
Superficial thrombophlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT02448771/Prot_SAP_000.pdf